CLINICAL TRIAL: NCT05195398
Title: TDCS to Improve Post-Stroke Cognitive Impairment
Acronym: TIPSCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland, College Park (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00315010
Record Dates: First submitted 2022-01-04; First posted 2022-01-19 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Stroke Sequelae; Cognitive Impairment
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to 15- 30 minute sessions of A-tDCS + CCT versus sham-intervention + CCT over a 5 week period
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A-tDCS (Experimental): Participants randomized to tDCS will undergo 15- 30 minute sessions over 5 weeks of A-tDCS to the ipsilesional frontoparietal cortex while participating in computerized cognitive therapy (CCT).
  Interventions: Device: Anodal transcranial Direct Current Stimulation (A-tDCS)
- Sham Intervention (Active Comparator): Participants randomized to sham will undergo 15- 30 minute sessions over 5 weeks of a sham-intervention, also applied to the ipsilesional frontoparietal cortex, while participating in computerized cognitive therapy (CCT).
  Interventions: Device: Sham Intervention

INTERVENTIONS:
Device: Anodal transcranial Direct Current Stimulation (A-tDCS) — Participants randomized to tDCS will undergo 5 weeks of A-tDCS + CCT.
  Other Names: Computerized Cognitive Therapy (CCT)
  Arms: A-tDCS
Device: Sham Intervention — Participants randomized to sham-intervention will undergo 5 weeks of sham + CCT.
  Other Names: Computerized Cognitive Therapy (CCT)
  Arms: Sham Intervention

SUMMARY:
The investigators will conduct a randomized, double-blinded, sham-controlled trial of approximately 60 patients with minor stroke and post-stroke mild cognitive impairment (psMCI). Participants will be individually randomized on enrollment using a random number generator to treatment with anodal tDCS + computerized cognitive treatment (CCT) versus sham + CCT (approximately 30 patients in each arm). Clinical evaluation including assessment of cognition will be performed pre- and post-intervention by individuals on the study team blinded to the participant's intervention. Participants will also undergo functional neuroimaging with magnetoencephalography (MEG) pre- and post-intervention (1, 3, and 6 months post-stroke to evaluate for initial and longer-term effects of treatment on cerebral activation patterns and functional connectivity). Neuroimaging and clinical outcomes will be assessed to determine the effect of tDCS versus sham + CCT on psMCI.

DETAILED DESCRIPTION:
Vascular cognitive impairment, ranging from vascular mild cognitive impairment to vascular dementia, is a leading cause of progressive cognitive dysfunction second only to Alzheimer Disease. While the accumulation of ischemic infarcts or a large cortical stroke can result in permanent cognitive dysfunction, a single small stroke can also result in disabling impairment. The investigators have shown that small lesions, regardless of the location, result in acute cognitive decline. Similar to those with progressive vascular cognitive impairment, post-stroke MCI (psMCI) patients display slowed reaction times and dysfunction across multiple cognitive domains. Many significantly recover over the first 6 months. However, the heterogenous recovery and uncertainty regarding prognosis can lead to major life changes, such as early retirement or selling of homes, that substantially impact quality of life.

Magnetoencephalography (MEG) recordings in those with psMCI show temporal dispersion consistent with generalized disruption of cognitive networks during resting state, irrespective of lesion location. Evaluation of frequency spectra show bilaterally decreased beta power in the frontoparietal lobes correlating with impaired reaction times. Functional connectivity analyses at 6 months demonstrate increased inter-hemispheric connections that may explain or reflect a patient's improvement. It is currently unknown whether specific cognitive networks are involved, though based on the pattern of clinical deficits it would be reasonable to hypothesize that the frontoparietal network, responsible for executive function and higher level cognitive tasks, is disrupted to a greater extent than the limbic, responsible for emotion and memory. Neural modulation with transcranial direct current stimulation (tDCS) increases the likelihood of neural firing, strengthening connectivity by promoting long-term potentiation and facilitating task performance. As anodal tDCS only induces the firing of neurons near threshold, it follows that it is most effective and longest acting when paired with a task that engages focal activation. This is best seen in patients with aphasia undergoing speech-language therapy.

In this study, the investigators will determine the utility of A-tDCS in conjunction with computerized cognitive therapy (CCT) to treat psMCI. The investigators will recruit approximately 60 patients with subacute minor stroke and randomize the patients to A-tDCS administered over the ipsilesional frontoparietal cortex versus sham plus 15 sessions of cognitive therapy using a widely used online platform focused most on executive functioning and processing speed based on the investigators' preliminary work targeting deficits most specific to those with psMCI. The investigators hypothesize that tDCS will augment both generalized connectivity as well as the connectivity of specific networks targeted during training (most notably the frontoparietal) and that patients will show increased clinical improvement acutely after therapy that will last for months after treatment.

Along with clinical evaluation, the investigators will use MEG to evaluate cerebral activation patterns and connectivity pre- (1 month post-infarct) and post- (3 and 6 months post-infarct) intervention. The investigators will collect longitudinal MEG and clinical data through a multicenter collaboration of experts in the fields of stroke, dementia, and functional neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) presenting with neurological symptoms due to acute ischemic stroke (symptom onset within the week prior to admission).
2. Evidence on brain MRI of acute ischemic stroke (imaging negative strokes and TIAs will be excluded).
3. Native English speaker (by self-report) prior to stroke.
4. NIHSS <8 at initial follow-up visit (approximately 30 days post-stroke).
5. mRS 0-2 at initial follow-up visit.

Exclusion Criteria:

1. Primary intracerebral hemorrhage- as evidenced by blood on head CT or MRI.
2. Presence of proximal large vessel occlusion.
3. Cortical exam findings including aphasia or neglect.
4. Prior report or history of dementia or undertreated psychiatric illness.
5. Uncorrected hearing or visual loss.
6. Inability to attend treatment or follow-up sessions.
7. Inability to travel to College Park (UMD) for MEG recording sessions.
8. Presence of any of the following that would lead to significant artifact on MEG: cardiac pacemaker, intracranial clips, metal implants or external clips within 10mm of the head, metal implants in the eyes (unlikely given that all patients will have an MRI and criteria are similar).
9. Claustrophobia, obesity, and/or any other reason leading to difficulty staying in the MEG machine for up to 1 hour.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition as assessed by our Cognitive Battery | Administered at 1, 3, and 6 month post-stroke visits
  Our cognitive battery was designed to efficiently evaluate for psMCI. It combines the Montreal Cognitive Assessment, Grooved Pegboard, Hopkins Verbal Learning Test, Brief Visuospatial Memory Test, Delis-Kaplan Executive Function System, and Symbol Digit Modalities Test. T scores are averaged across tasks and calculated for the following cognitive domains: verbal memory, spatial memory, processing speed, motor speed, executive function, and global cognition.
Change in Functional Connectivity as assessed by MEG | Administered at 1, 3, and 6 month post-stroke visits
  Participants will undergo an MEG evaluating global functional connectivity: 1) during resting state, and 2) during completion of a visual task. Connectivity will also be evaluated within the following specific cognitive networks: frontoparietal (executive) and limbic (memory)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth B Marsh, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Results in aggregate will be posted; however, de-identified individual participant data will be made available to other investigators and potential collaborators upon reasonable request of the PI.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: One year following completion of data collection and publication of results.

REFERENCES:
- [Background] Marsh EB, Brodbeck C, Llinas RH, Mallick D, Kulasingham JP, Simon JZ, Llinas RR. Poststroke acute dysexecutive syndrome, a disorder resulting from minor stroke due to disruption of network dynamics. Proc Natl Acad Sci U S A. 2020 Dec 29;117(52):33578-33585. doi: 10.1073/pnas.2013231117. Epub 2020 Dec 14. PMID 33318200
- [Background] Marsh EB, Lawrence E, Hillis AE, Chen K, Gottesman RF, Llinas RH. Pre-stroke employment results in better patient-reported outcomes after minor stroke: Short title: Functional outcomes after minor stroke. Clin Neurol Neurosurg. 2018 Feb;165:38-42. doi: 10.1016/j.clineuro.2017.12.020. Epub 2017 Dec 27. PMID 29306185
- [Background] Sharma R, Mallick D, Llinas RH, Marsh EB. Early Post-stroke Cognition: In-hospital Predictors and the Association With Functional Outcome. Front Neurol. 2020 Dec 23;11:613607. doi: 10.3389/fneur.2020.613607. eCollection 2020. PMID 33424761
- See also: Marsh Lab website — http://www.marshlab.org